CLINICAL TRIAL: NCT04484363
Title: Expanded Access Program: Pevonedistat (in Combination With Azacitidine) for the First-line Treatment of Higher Risk Myelodysplastic Syndromes
Brief Title: Expanded Access Program With Pevonedistat (Given With Azacitidine) for Adults With Higher-risk Myelodysplastic Syndromes
Status: No longer available | Type: Expanded Access
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Pevonedistat-5005
Record Dates: First submitted 2020-07-22; First posted 2020-07-23 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Drug Therapy
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — pevonedistat; Azacitidine

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Pevonedistat — Pevonedistat 20 milligram per square meter (mg/m^2), intravenous infusion, on Days 1, 3, and 5 of repeated 28-day cycles.
Drug: Azacitidine — Azacitidine 75 mg/m^2, intravenous or subcutaneous infusion, on Days 1 to 5, Days 8 and 9 of repeated 28-day cycles or Days 1 through 7 of repeated 28-day cycles.

SUMMARY:
Participants in the expanded access program are adults with higher-risk myelodysplastic syndromes who have no other treatment options available.

The main aim of this program is to allow participants to have access to pevonedistat before FDA approval.

This program will take place in the United States.

DETAILED DESCRIPTION:
This is an expanded access program in which the drug being tested is called pevonedistat, which is used in combination with azcitidine. This study will provide expanded access of pevonedistat (in combination with azacitidine) for the first-line treatment to participants with HR-MDS and option of real world data (RWD) collection for the benefit of future participants.

All participants will receive azacitidine via intravenous or subcutaneous route in combination with pevonedistat intravenous infusion.

This multi-center trial will be conducted in the United States. Participant will continue treatment until benefit is no longer derived from the treatment (that is, until disease progression, or treatment is no longer tolerable), the benefit-risk no longer favors the individual, an appropriate alternative therapy becomes available, the participant chooses to discontinue the treatment, or pevonedistat becomes commercially available.

ELIGIBILITY:
Inclusion Criteria:

1. Has morphologically confirmed diagnosis of MDS.
2. With MDS have one of the following Prognostic Risk Categories, based on the Revised International Prognostic Scoring System (IPSS-R)

   * Very high (greater than [>] 6 points).
   * High (>4.5-6 points).
   * Intermediate (>3-4.5 points): a participant determined to be in the Intermediate Prognostic Risk Category is only allowable in the setting of greater than or equal to (>=) 5 percent (%) bone marrow myeloblasts.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2.
4. Has never been treated with Azacitidine, or, has been treated with Azacitidine, two or fewer cycles of Azacitidine have been administered, and has not relapsed while being treated with Azacitidine or failed Azacitidine treatment.

Exclusion Criteria:

1. Has previous treatment for HR MDS with chemotherapy or other antineoplastic agents including hypomethylating agent (HMAs) such as decitabine or more than two cycles of azacitidine.

   • Previous treatment with lenalidomide is permitted, except that lenalidomide may not be given within 8 weeks of first dose of drug.
2. Has acute promyelocytic leukemia as diagnosed by morphologic examination of bone marrow, by fluorescent in situ hybridization or cytogenetics of peripheral blood or bone marrow, or by other accepted analysis.
3. Has either clinical evidence of or history of central nervous system involvement by acute myelogenous leukemia (AML).
4. Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia.
5. Has prothrombin time (PT) or activated partial thromboplastin time (aPTT) >1.5*upper limit of normal (ULN) or active uncontrolled coagulopathy or bleeding disorder. Participants therapeutically anticoagulated with warfarin, direct thrombin inhibitors, direct factor Xa inhibitors, or heparin are excluded from enrollment.
6. Has known hepatitis B surface antigen seropositivity, or known or suspected active hepatitis C infection. Note: Participants who have isolated positive hepatitis B core antibody (that is, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Participants who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
7. Has known hepatic cirrhosis or severe preexisting hepatic impairment.
8. Has known cardiopulmonary disease defined as unstable angina, clinically significant arrhythmia, congestive heart failure (New York Heart Association Class III or IV), and/or myocardial infarction within 6 months before first dose, or severe pulmonary hypertension.
9. Has treatment with strong cytochrome P 3A (CYP3A) inducers within 14 days before the first dose of pevonedistat.

   .

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a3be